CLINICAL TRIAL: NCT04648696
Title: Safety and Outcomes Associated With Continuous Versus Intermittent Infusion Vancomycin in Outpatient Parenteral Antibiotic Therapy: a Prospective, Randomized Trial
Brief Title: Safety and Outcomes Associated With Continuous Versus Intermittent Infusion Vancomycin
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was closed due to slow enrollment.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00069815
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2022-09

CONDITIONS: Infection
Keywords: infusion therapy; continuous infusions; nephrotoxicity; outpatient parenteral antibiotic therapy; vancomycin
MeSH Terms: conditions — Infections | interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: To assess the risk of vancomycin-associated nephrotoxicity and outcomes associated with continuous infusions (CI) versus II dosing in the outpatient parenteral antibiotic therapy (OPAT) setting
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- continuous infusions (CI) group (Active Comparator): CI group will have their total daily cumulative dose of vancomycin converted to a 24-hour intravenous infusion upon discharge
  Interventions: Drug: Vancomycin CI
- Intermittent infusion (II) group (Active Comparator): Inpatient study candidates that are randomized to the II group will continue their current intravenous dosing upon discharge
  Interventions: Drug: Vancomycin II

INTERVENTIONS:
Drug: Vancomycin CI — The CI group will have their total daily cumulative dose of vancomycin converted to a 24-hour intravenous infusion upon discharge - the CI will begin with the first scheduled OPAT dose of vancomycin
  Other Names: glycopeptide antibiotic
  Arms: continuous infusions (CI) group
Drug: Vancomycin II — Study candidates that are randomized to the II group will continue their current intravenous dosing upon discharge
  Other Names: glycopeptide antibiotic
  Arms: Intermittent infusion (II) group

SUMMARY:
Evaluate the safety and outcomes associated between the two treatment modalities

DETAILED DESCRIPTION:
Assess the risk of vancomycin-associated nephrotoxicity and outcomes associated with continuous infusions (CI) versus II dosing in the outpatient parenteral antibiotic therapy (OPAT) setting

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at least 18 years of age
* Receiving Wake Forest Baptist Health Outpatient parenteral antimicrobial therapy (OPAT) services
* Will receive vancomycin therapy from Wake Forest Baptist Health Specialty Home Infusion Pharmacy
* Planned therapy with vancomycin in the outpatient setting for at least 2 weeks in duration
* Prescribed vancomycin with a frequency of either every 12 hours or every 8 hours dosing at the time of enrollment

Exclusion Criteria:

* Presence of diseases or conditions known to affect the pharmacokinetics of vancomycin: Pregnancy/Ascites/Burn injury/Cystic fibrosis /Weight greater-than or equal-to 150 kg
* Pre-existing leukopenia: White Blood Cell (WBC) < 4,000 x 103 cells/µL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Williamson, PharmD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 Subject Screen Failed who never received study treatment
Groups:
- Continuous Infusions (CI) Group: continuous infusions (CI) group will have their total daily cumulative dose of vancomycin converted to a 24-hour intravenous infusion upon discharge
  Vancomycin CI: The CI group will have their total daily cumulative dose of vancomycin converted to a 24-hour intravenous infusion upon discharge - the CI will begin with the first scheduled OPAT dose of vancomycin
Period: Overall Study
Arm/Group | Continuous Infusions (CI) Group | Intermittent Infusion (II) Group
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Infusions (CI) Group | Intermittent Infusion (II) Group | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Full Range); unit: years] | 44 [24 to 62] | 57 [46 to 63] | 49 [24 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Nephrotoxicity in Subjects
Description: Number of Subjects with any increase in Serum creatinine by 50% from baseline, an increase in Scr by 0.5 mg/dL, or an increase in Scr by 0.3 mg/dL on two consecutive measurements
Time Frame: week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Infusions (CI) Group | Intermittent Infusion (II) Group
Number analyzed (Participants) | 4 | 3
Participants | 0 | 1

2. Secondary Outcome: Number of Leukopenia in Subjects
Description: Number of Subjects with White Blood Cell (WBC) < 4,000 x 103 cells/µL
Time Frame: week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Infusions (CI) Group | Intermittent Infusion (II) Group
Number analyzed (Participants) | 4 | 3
Participants | 1 | 0

3. Secondary Outcome: Number of Infusion-related Reactions
Description: Flushing/Erythema /Rash/Red Man Syndrome
Time Frame: week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Infusions (CI) Group | Intermittent Infusion (II) Group
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

4. Secondary Outcome: Number of Serum Vancomycin Measurements Within Therapeutic Range
Description: Number of Serum Vancomycin Measurements Within Therapeutic Range If inpatient dose was determined by AUC monitoring: A vancomycin trough that is within 3.0 mcg/mL of the trough that correlated with a therapeutic AUC based on inpatient monitoring - If inpatient dose was not determined by AUC monitoring or vancomycin was initiated as outpatient: A vancomycin trough of 10.0 - 20.0 mcg/mL
Time Frame: week 8
Measure: Number; unit: Number of Blood Draws
Units Other Than Participants: Number of blood draws
Arm/Group | Continuous Infusions (CI) Group | Intermittent Infusion (II) Group
Number analyzed (Participants) | 4 | 3
Number analyzed (Number of blood draws) | 15 | 8
Number of Blood Draws | 9 | 2

5. Secondary Outcome: Number of Participants With Resolutions of Symptoms Associated With the Infection
Description: Number of Subjects without need for additional induction therapy beyond the planned end date
Time Frame: week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Infusions (CI) Group | Intermittent Infusion (II) Group
Number analyzed (Participants) | 4 | 3
Participants | 3 | 1

6. Secondary Outcome: Number of Participants With Treatment Failures
Description: Number of Participants with Persistence, new onset, or worsening local or systemic signs and symptoms of infection
Time Frame: week 21
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Infusions (CI) Group | Intermittent Infusion (II) Group
Number analyzed (Participants) | 4 | 3
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: up to 21 weeks
Arm/Group | Continuous Infusions (CI) Group | Intermittent Infusion (II) Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 1/4 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Infusions (CI) Group (N=4) | Intermittent Infusion (II) Group (N=3)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — an abnormal reduction of circulating white blood cells, especially the granulocytes
hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
nephrotoxicity (Renal and urinary disorders) | 0 (0) | 1 (1) — kidneys are damaged by a drug, chemical or toxin, resulting in possible chronic kidney disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT04648696/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT04648696/ICF_002.pdf